CLINICAL TRIAL: NCT03903107
Title: Fluoroless Conduction System Pacing Utilizing Electro-Anatomic Mapping Versus Conventional Implantation: The Fluoroless- CSP Trial
Brief Title: The Fluoroless-CSP Trial Using Electroanatomic Mapping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18090701
Record Dates: First submitted 2018-10-31; First posted 2019-04-04 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Sinus Node Dysfunction; Heart Block AV; LBBB; Heart Failure, Systolic
MeSH Terms: conditions — Sick Sinus Syndrome; Atrioventricular Block; Heart Failure, Systolic

STUDY DESIGN:
Intervention Model Description: CSP can be achieved successfully and safely utilizing electro-anatomic mapping (EAM) with the CARTO 3mapping system
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Conduction System Pacing(CSP) using fluoroscopy (Placebo Comparator): Subjects in this arm will receive Conduction System Pacing(CSP) using conventional fluoroscopy technique.
  Interventions: Procedure: Conventional fluoroscopy guided Conduction System Pacing(CSP)
- Fluoroless Conduction System Pacing(CSP) utilizing EAM with the CARTO 3 mapping system (Experimental): Subjects in this arm will receive Conduction System Pacing(CSP) utilizing electroanatomic mapping system to eliminate or minimize fluoroscopic exposure.
  Interventions: Procedure: Electroanatomic Mapping (Fluoroless) guided Conduction System Pacing(CSP)

INTERVENTIONS:
Procedure: Conventional fluoroscopy guided Conduction System Pacing(CSP) — conventional standard approach Conduction System Pacing(CSP) using fluoroscopy
  Arms: Conventional Conduction System Pacing(CSP) using fluoroscopy
Procedure: Electroanatomic Mapping (Fluoroless) guided Conduction System Pacing(CSP) — Conduction System Pacing(CSP) using electroanatomic mapping system with no or minimal fluoroscopy
  Arms: Fluoroless Conduction System Pacing(CSP) utilizing EAM with the CARTO 3 mapping system

SUMMARY:
The goal of this study is to assess the feasibility, accuracy and safety of performing fluoroless (or low fluoro) conduction system pacing utilizing electro-anatomic mapping (EAM) with the CARTO 3 mapping system (Biosense Webster Inc, Irvine, CA) in comparison to a group of patients undergoing conventional conduction system pacing (CSP) Implants.

DETAILED DESCRIPTION:
The goal of this study is to assess the feasibility, accuracy and safety of performing fluoroless (or low fluoro) conduction system pacing utilizing electro-anatomic mapping (EAM) with the CARTO 3 mapping system (Biosense Webster Inc, Irvine, CA) in comparison to a group of patients undergoing conventional conduction system pacing (CSP) Implants.

In this study, we plan to randomize patients to fluoroscopy guided CSP vs 3D mapping guided CSP implants with low/zero fluoroscopy. The study with assess if 3D EAM guided implants can be performed successfully and without any significant increase in device implant related complications.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Indication for Permanent Pacemaker implantation or implantation of Cardiac Resynchronization Therapy Device

Exclusion Criteria:

* Existing cardiac device including Pacemaker or Cardiac Resynchronization Therapy device
* Inability of patient capacity to provide consent for themselves either due to medical or psychiatric comorbidity
* Pregnancy
* Difficulty with follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Success of achieving CSP | Intra-procedure
  Feasibility of achieving a successful CSP implant at the His Bundle or Left Bundle branch with low or zero Fluoroscopy. This will result in low to no fluoroscopy exposure for both the subject and the operator, as well as shorter procedure times.This will be documented during procedure.

SECONDARY OUTCOMES:
Total radiation exposure time during procedure | Intra-procedure
  Total radiation exposure during procedure time will be documented at the total time the patient is exposed to fluoroscopy during the procedure. This will will be tracked and documented as total fluoroscopy duration, His lead Fluoroscopy duration and DAP. The total amounts of procedural fluoroscopy exposure will be compared between the two treatment arms.
Procedure-related complications | 30 days post procedure
  The study team will review medical history of enrolled subjects for any adverse event experienced post-procedurally. All adverse events will be reviewed by PI for determination as to whether "procedure-related" or not.
Need for His Lead revisions | for a period of 6 months post procedure
  The study team will track the device follow-up data for a duration of 3 months post device implant. Any patients with > 2V increase in His Lead capture threshold from baseline and need for ventricular pacing will undergo a lead revision.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sharma PS, Huang HD, Trohman RG, Naperkowski A, Ellenbogen KA, Vijayaraman P. Low Fluoroscopy Permanent His Bundle Pacing Using Electroanatomic Mapping: A Feasibility Study. Circ Arrhythm Electrophysiol. 2019 Feb;12(2):e006967. doi: 10.1161/CIRCEP.118.006967. PMID 30704289